CLINICAL TRIAL: NCT06785597
Title: EpigenOMic Determinants of the Neuroendocrine Phenotype As Biomarkers for Noninvasive Diagnosis of Neuroendocrine Neoplasms
Brief Title: EpigenOMic Determinants of the Neuroendocrine Phenotype As Biomarkers for Neuroendocrine Neoplasms
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Sponsor
Other Study IDs: L2-154
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-08

CONDITIONS: Mixed Neuroendocrine-Non Neuroendocrine Neoplasm; Neuroendocrine Neoplasm
Keywords: global molecular profiling; neuroendocrine phenotype; biomarker; epigenomic determinant
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples; surgical/bioptic samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neuroendocrine neoplasm case: patient with histologically confirmed neuroendocrine neoplasm and onfirmed Mixed Neuroendocrine-non neuroendocrine neoplasm with each component > 30%) and high-grade Neuroendocrine Carcinomas
- Non-neuroendocrine neoplasm control: patient with histologically confirmed non-neuroendocrine gastrointestinal tumors (including gastric, pancreatic, colorectal, small intestine).

SUMMARY:
For GEP mixed neuroendocrine (NE) non-neuroendocrine neoplasms (MiNENs) a key issue affecting prognosis is sometimes the difficulty in obtaining a timely diagnosis, as the NE component is often localized in deeper anatomical locations and/or becomes prevalent over time. The tissue material of biopsies may be not enough to define the NE component when this is particularly small and this could impact on therapeutic decision. Furthermore GEP NENs need to be characterized for potentially druggable biomarkers and liquid biopsy has clear advantage to the solid one to this aim. Here, we will exploit epigenetic differences characterizing NE tumors to build a DNA methylation-based liquid biopsy assay able to detect circulating tumor DNA of NE derivation, to enable the non-invasive diagnosis and monitoring of GEP-MiNENs.

DETAILED DESCRIPTION:
GEP-NENs are a heterogeneous group of diseases that encompasses relatively indolent and more aggressive tumors, sometimes with mixed exocrine/endocrine components (MINENs). Due to persistent uncertainties in diagnosis and treatment, prognosis of the mixed and more aggressive forms remains poor. Non-invasive tests would enable timely identification and monitoring over time. A better understanding of their biology and of the phenotypic differentiation process may pave the way for novel therapies. Differentiation follows, and can be inferred from, changes in the epigenetic landscape that shape transcriptional programs. Among epigenetic markers, DNA methylation is particularly well suited for non-invasive detection as it can be measured in circulating tumor DNA (ctDNA). New technologies like Oxford Nanopore Technologies (ONT) enable simultaneous analysis of DNA sequence and methylation, as we recently showed by Magi et al Nat Comms Biol 2022. Previous studies identified distinct neuroendocrine epi-transcriptomic landscapes but were conducted on tumor specimens (Yachida et al Cancer Discov 2022), impeding the discrimination of signals specifically generated within neuroendocrine tumor cells from the noise due to surrounding nontumoral or exocrine tumoral cells. This is now potentially solved by methods allowing single-cell sequencing directly from frozen or paraffin-embedded patient samples.

The main expected outcome is the development of a novel liquid biopsy assay for the detection and monitoring of GEP-NENs and MiNENs. To this end, we will exploit the ability of Oxford Nanopore Technologies (ONT) sequencing to simultaneously yield sequencing and methylated DNA profiles. Importantly, assessment of cell of origin from ctDNA requires the comparison of methylation and fragmentomics signals with previously generated maps of reference cells and tissues (Katsman et al 2022 Genome Biology). For rare tumors like NENs, these maps are not available in the literature; the few studies that have characterized the epigenomic features of NENs are likely contaminated by the surrounding stroma, so epigenetic signals (including both DNA methylation and tumor-specific transcription factor binding sites, essential for fragmentomics) may be uninformative for detection in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed diagnosis of NEC/MINEN amenable to surgery with radical intent
* Patient with histologically confirmed diagnosis of NET amenable to surgery with radical intent
* Patient with metastatic NET/NEC, amenable to biopsy or surgery, including palliative intent
* Patient histologically confirmed non-NEN histotype:

  1. Colorectal carcinoma
  2. Small intestine carcinoma
  3. Gastric or oesophageal carcinoma
  4. Pancreatic ductal adenocarcinoma
  5. Metastasectomy from any non-NEN GI carcinoma

Exclusion Criteria:

* Grading G1 and G2 <=10% Ki67
* Presence of concomitant neoplasm (within 3 years)
* Concomitant major haematological alteration
* Concomitant major organ dysfunction (e.g. G3/4 liver or kidney failure)
* Ongoing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GEP-NENs, aiming to collect adequate material and for a formal clinical to establish sensitivity and specificity of the assay in a clinically meaningful scenario.
  Due to the relative rarity of the disease compared to non-NENs we will not enroll a consecutive population, but we will set up a case-control study:
  * Cases: patients with resectable, histologically confirmed NENs
  * Controls: patients with resectable, histologically confirmed non-neuroendocrine gastrointestinal tumors (including gastric, pancreatic, colorectal, small intestine).
  Patients will be enrolled as cases or controls based on their pre-surgical diagnostic biopsy but will be definitively allocated in the case or control group based on their post-surgery full histological examination.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Develop a circulating methDNA/fragmentomics diagnostic assay | 2 years
  Epigenetic differences characterizing neuroendocrine tumors will be exploited to build a DNA methylation-based liquid biopsy assay able to detect circulating tumor DNA of neuroendocrine derivation, to enable the non-invasive diagnosis and monitoring of GEP-MiNENs.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Fazio, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy